CLINICAL TRIAL: NCT00791635
Title: Longitudinal Evaluation of Women Undergoing Pelvic Exenteration for Treatment of Gynecologic Malignancy
Brief Title: Longitudinal Evaluation of Women Undergoing Pelvic Surgery for the Treatment of Gynecologic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0095; NCI-2020-07746 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0095 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cervical Carcinoma; Endometrial Carcinoma; Malignant Female Reproductive System Neoplasm; Vaginal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaires): RETROSPECTIVE PORTION: Patients who have undergone pelvic exenteration complete one set of QOL questionnaires.
  PROSPECTIVE PORTION: Patients undergoing pelvic exenteration complete questionnaires over 20-40 minutes within 2 weeks before surgery, and at 4-12 weeks, 6 months, and 1, 2, 3, 4, 5, and 10 years after surgery regarding feelings, abilities, depression, coping, social support, sexual function and body image. Patients with cervical cancer may complete 1 additional questionnaire during each of these visits.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
The study investigates whether certain characteristics of gynecological cancer can help researchers predict how well a patient recovers from surgery to remove the lower colon, rectum, and bladder, and create openings through which urine and stool are passed out of the body (pelvic exenteration). Comparing the types of surgery completed and procedures used may help researchers to determine which are most effective and safe in patients with a history of gynecologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the types of complications experienced by women who undergo pelvic exenteration at University of Texas (UT) MD Anderson Cancer Center.

II. To determine whether the number of complications experienced by women who undergo pelvic exenteration at UT MD Anderson Cancer Center differ by vaginal and bladder reconstruction types.

SECONDARY OBJECTIVES:

I. To evaluate pathologic predictors of recurrence including histology, size of tumor, and distance of closest margin.

II. To longitudinally assess quality of life, sexual functioning, and symptoms in women who have undergone pelvic exenteration for gynecologic malignancies.

III. To assess the impact of certain preoperative factors (albumin, electrolyte levels, body mass index) on the occurrence of post-operative complications.

IV. To determine if preoperative positron emission tomography (PET)/computed tomography (CT) correlates with pathologic findings at the time of surgery.

V. To calculate time to recurrence, overall survival, and disease-free survival of patients who undergo pelvic exenteration and correlate to key demographic, clinical, and pathologic factors.

OUTLINE:

RETROSPECTIVE PORTION: Patients who have undergone pelvic exenteration complete one set of quality of life (QOL) questionnaires.

PROSPECTIVE PORTION: Patients undergoing pelvic exenteration complete questionnaires over 20-40 minutes within 2 weeks before surgery, and at 4-12 weeks, 6 months, and 1, 2, 3, 4, 5, and 10 years after surgery regarding feelings, abilities, depression, coping, social support, sexual function and body image. Patients with cervical cancer may complete 1 additional questionnaire during each of these visits.

Patients who undergo surgery are followed up every 3 months for the first 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of gynecologic malignancy, including cervical, endometrial, vulvar, or vaginal carcinoma of any histology
* Women who have undergone a pelvic exenteration after January 1993 or who are being offered a pelvic exenteration for treatment of their gynecologic malignancy
* Patients must be suitable candidates for surgery (in case of prospective collection)
* Patients who have signed an approved informed consent
* Patients with a prior malignancy allowed if > 3 years previous with no current evidence of disease
* Women must be able to read and write in either Spanish or English

Exclusion Criteria:

* Patients with contraindications to surgery
* Patients unwilling or unable to complete self-administered questionnaires
* Patients who do not read or speak English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a history of gynecologic malignancy who have undergone or are being offered a pelvic exenteration
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2008-07-11 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of surgical complications | 4 years
  Will determine whether the number of surgical complications varies by vaginal and bladder reconstruction type.
Short-term and long-term complications | 4 years
  Will calculate incidence with exact 95% confidence intervals, and will calculate summary statistics. Will create the statistics using both cohorts of patients together. Will also do this separately by cohort and by vaginal reconstruction type as well as by bladder reconstruction type. A Wilcoxon rank-sum test will be used to determine whether there is a difference in number of complications by vaginal reconstruction type and by bladder reconstruction type. This will be conducted separately for each cohort. Finally, will create a Poisson regression model using both cohorts of patients with terms for cohort, vaginal reconstruction type and bladder reconstruction type as well as certain preoperative factors (albumin, electrolyte levels, body mass index) that might be predictive of number of complications.
Quality of life | Up to 5 years
  Will summarize composite scores of the quality of life surveys by time from exenteration. This will be done separately for the retrospectively recruited patients and the prospectively recruited patients. Will also summarize information by year of surgery. To determine how quality of life changes over time, will create longitudinal models for each survey instrument given to the women. The two cohorts of women will initially be analyzed separately. A second model will be created using all patients that has terms for cohort, vaginal reconstruction type and bladder reconstruction type to determine whether these terms have an effect upon quality of life.
Recurrence | Up to 5 years
  Will calculate median time to recurrence in patients who undergo pelvic exenteration. Will use log-rank tests and construct proportional hazards models to evaluate pathologic predictors of recurrence such as histology, size of tumor, and distance of closest margin.
Overall survival | Up to 5 years
  Will calculate overall survival of patients who undergo pelvic exenteration. Will use log-rank tests and construct proportional hazards models to evaluate pathologic predictors of survival such as histology, size of tumor, and distance of closest margin.
Disease-free survival | Up to 5 years
  Will calculate disease-free survival of patients who undergo pelvic exenteration. Will use log-rank tests and construct proportional hazards models to evaluate pathologic predictors of survival such as histology, size of tumor, and distance of closest margin.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela T Soliman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org